CLINICAL TRIAL: NCT02781285
Title: Effect Study of Clinical Outcomes of Traditional Chinese Medicine to Advanced Gastric Cancer by Propensity Score Through Registration
Brief Title: Effect Study of Clinical Outcomes of Traditional Chinese Medicine to Advanced Gastric Cancer by Propensity Score
Acronym: ESCOTCMAGCPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); RenJi Hospital (Other); Fudan University (Other); ShuGuang Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Ruijin Hospital (Other); Yunnan Provinical Hospital of Traditional Chinese Medicine (Other); Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other); Shaanxi Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: LONGHUA-2016-SH
Record Dates: First submitted 2016-05-15; First posted 2016-05-24 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Gastric Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1group one: patients with standard TCM diagnosis and treatment of gastric cancer
- 2 group two: patients take Chinese Medicine but not with standard TCM diagnosis and treatment of gastric cancer
- 3group three: patients take no Chinese Medicine

SUMMARY:
The researching subject is aimed to obtain the clinical evidences (including real benefits， risks ,etc. ) of traditional Chinese medicine in the treatment of advanced gastric cancer by compared with the outcomes that not accept the traditional Chinese medicine. the subject acquires these clinical practices by using the methods of multicenter、persisting registry (the real world researching technology ) and propensity score.

DETAILED DESCRIPTION:
The purpose of this project is to further evaluate the role of traditional Chinese medicine in the treatment of advanced gastric cancer through clinical registration along with real world study.

The patients who suffer from advanced gastric cancer often have a very short time survival . Their total survival time is only 4.3 months after the best supportive care. At present palliative chemotherapy is still the main method for advanced gastric cancer .

In recent years, the results of international multi center phase III clinical trial show that the patients with combination chemotherapy have 8.6 months to 13.0 months survival time.

In China, the clinical curative effect of traditional Chinese medicine in the treatment of advanced gastric cancer has been part of affirmation. Some reports with large samples of clinical research show that the Traditional Chinese Medicine may prolong the survival and improve the quality of life in patients with advanced gastric cancer.

Real World Study emphasizes in epidemiological theories, clinical observational study, cross-sectional study and cohort study. The observational study of registry (registry study in clinical practice) is particularly widely used.

Clinical practice of traditional Chinese medicine in the treatment of advanced gastric cancer often relies on the accumulation of years of medical experiences and sometimes new treatment measures. There must be some objective evidences that with reasonable design, rigorous process, scientific statistics to evaluate the value of traditional Chinese medicine intervention in the comprehensive treatment of advanced gastric cancer patients in order to meet the needs of clinical practice and medical development in China.

ELIGIBILITY:
Inclusion Criteria:

* gastric adenocarcinoma without operation or recurrence after operation or metastasis
* diagnosed within three months
* KPS score≥60
* expected survival time was above 3 months
* HB ≥80g/L 、WBC≥4.0×109/L、 N ≥2.0×109/L 、PLA ≥80×109/L
* normal function with heart 、kidney and liver

Exclusion Criteria:

* not gastric adenocarcinoma
* simultaneous diagnosis with other malignant tumor
* participate in clinical trials of new drugs not listed in China
* combined with myocardial infarction, cerebral infarction, severe liver and kidney dysfunction, postoperative severe complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both: both female and male participants are being studied
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2014-12 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The influences of traditional Chinese medicine standardized treatment on the overall survival (OS) of patients with advanced gastric cancer by the method of Propensity Score. | two years
  Two years of continuous observation after the initial diagnosis of advanced gastric cancer with 725 cases .

SECONDARY OUTCOMES:
The influences of traditional Chinese medicine treatment but with standardization scheme on the overall survival (OS) of patients with advanced gastric cancer by the method of Propensity Score. | two years
  Two years of continuous observation after the initial diagnosis of advanced gastric cancer with 375 cases.
The influences of Western Medicine treatment mainly by chemotherapy on the overall survival (OS) of patients with advanced gastric cancer by the method of Propensity Score. | two years
  Two years of continuous observation after the initial diagnosis of advanced gastric cancer with 400 cases.

CONTACTS AND LOCATIONS:
Overall Officials: zhao ai guang, Dr., Principal Investigator — Shanghai Longhua Hospital
Locations (1):
- Longhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Yilmaz U, Oztop I, Alacacioglu A, Yaren A, Tarhan O, Somali I. Irinotecan combined with infusional 5-fluorouracil and high-dose leucovorin for the treatment of advanced gastric carcinoma as the first-line chemotherapy. Chemotherapy. 2006;52(5):264-70. doi: 10.1159/000094769. Epub 2006 Jul 26. PMID 16873996
- [Derived] Cao ND, Zhu XH, Ma FQ, Xu Y, Dong JH, Qin MM, Liu TS, Zhu CC, Guo WJ, Ding HH, Guo YB, Liu LK, Song JJ, Wu JP, Cheng YL, Zeng L, Zhao AG. Chinese Medicine Prolongs Overall Survival of Chinese Patients with Advanced Gastric Cancer: Treatment Pattern and Survival Analysis of a 20-Year Real-World Study. Chin J Integr Med. 2024 Jun;30(6):489-498. doi: 10.1007/s11655-024-4107-8. Epub 2024 May 27. PMID 38801641